CLINICAL TRIAL: NCT05415137
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Intravenous Efzofitimod in Patients With Pulmonary Sarcoidosis
Brief Title: Efficacy and Safety of Intravenous Efzofitimod in Patients With Pulmonary Sarcoidosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Collaborators: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATYR1923-C-004
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Pulmonary Sarcoidosis; Sarcoidosis; Granuloma; Inflammation; Lymphoproliferative Disorders; Interstitial Lung Disease; Neuropilin-2; Steroids; Oral corticosteroids; Immunomodulatory; tRNA Synthetase; ATYR1923; KRP-R120; Efzofitimod; Fibrosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis; Granuloma; Inflammation; Lymphoproliferative Disorders; Lung Diseases, Interstitial; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efzofitimod 3 mg/kg (Experimental)
  Interventions: Drug: Efzofitimod 3 mg/kg
- Efzofitimod 5 mg/kg (Experimental)
  Interventions: Drug: Efzofitimod 5 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efzofitimod 3 mg/kg — EfzofitimodIV infusion every 4 weeks for a total of 12 doses
  Other Names: ATYR1923; KRP-R120
  Arms: Efzofitimod 3 mg/kg
Drug: Efzofitimod 5 mg/kg — EfzofitimodIV infusion every 4 weeks for a total of 12 doses
  Other Names: ATYR1923; KRP-R120
  Arms: Efzofitimod 5 mg/kg
Drug: Placebo — Placebo IV infusion every 4 weeks for a total of 12 doses
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, study comparing the efficacy and safety of intravenous (IV) efzofitimod 3 mg/kg and 5 mg/kg versus placebo after 48 weeks of treatment. This study will enroll adults with histologically confirmed pulmonary sarcoidosis receiving stable treatment with oral corticosteroid (OCS), with or without immunosuppressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of pulmonary sarcoidosis for at least 6 months, supported by the following evidence: documented histologically proven diagnosis of sarcoidosis by tissue biopsy and documented evidence of parenchymal lung involvement by historical radiological evidence
* Evidence of symptomatic pulmonary sarcoidosis, as demonstrated by the following criteria: Modified Medical Research Council (MRC) dyspnea scale grade of at least 1 and KSQ-Lung score ≤70
* Patients must be receiving treatment with OCS of ≥ 3 months at Day 1 with a starting dose between ≥ 7.5 and ≤ 25 mg/day ≥ 4 weeks prior to Day 1.
* Body weight ≥ 40 kg and < 160 kg

Exclusion Criteria:

* Treatment with > 1 immunosuppressant therapy
* Treatment with biological immunomodulators, such as tumor necrosis factor-alpha (TNF-α) inhibitors or antifibrotics or interleukin inhibitors
* Likelihood of significant pulmonary fibrosis as shown by any 1 or more of the following: High resolution CT fibrosis > 20% within the last 12 months; FVC percent predicted (FVCPP) < 50% and KSQ-Lung score < 30
* In the opinion of the investigator, clinically significant pulmonary hypertension
* Patients with active cardiac, neuro, or renal sarcoidosis requiring organ-specific therapy in the past 2 years
* Patients with cutaneous or ocular sarcoidosis, which in the opinion of the Investigator, are at risk for exacerbation, necessitating OCS rescue or other systemic therapy
* History of Addisonian symptoms that precluded previous OCS taper attempts
* Is an active, heavy smoker of tobacco/nicotine-containing products
* History of anti-synthetase syndrome or Jo-1 positive at Screening
* Patients with active tuberculosis or those currently undergoing treatment for tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean daily oral corticosteroid (OCS) dose at Week 48 | Baseline to Week 48

SECONDARY OUTCOMES:
Change from baseline in KSQ-Lung score at Week 48 | Baseline to Week 48
Steroid withdrawal rate | Baseline to Week 48
Change from baseline in absolute value of FVC at Week 48 | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carey, Study Director — aTyr Pharma, Inc.
Locations (82):
- United States (37):
  - aTyr Investigative Site, Birmingham, Alabama
  - aTyr Investigative Site, Phoenix, Arizona
  - aTyr Investigative Site, Los Angeles, California
  - aTyr Investigative Site, Sacramento, California
  - aTyr Investigative Site, Denver, Colorado
  - aTyr Investigative Site, Washington D.C., District of Columbia
  - aTyr Investigative Site, Gainesville, Florida
  - aTyr Investigative Site, Tampa, Florida
  - aTyr Investigative Site, Weston, Florida
  - aTyr Investigative Site, Atlanta, Georgia
  - aTyr Investigative Site, Chicago, Illinois
  - aTyr Investigative Site, Louisville, Kentucky
  - aTyr Investigative Site, New Orleans, Louisiana
  - aTyr Investigative Site, Baltimore, Maryland
  - aTyr Investigative Site, Boston, Massachusetts
  - aTyr Investigative Site, Ada, Michigan
  - aTyr Investigative Site, Detroit, Michigan
  - aTyr Investigative Site, Minneapolis, Minnesota
  - aTyr Investigative Site, Rochester, Minnesota
  - aTyr Investigative Site, Jackson, Mississippi
  - aTyr Investigative Site, St Louis, Missouri
  - aTyr Investigative Site, Albany, New York
  - aTyr Investigative Site, Middletown, New York
  - aTyr Investigative Site, Durham, North Carolina
  - aTyr Investigative Site, Greenville, North Carolina
  - aTyr Investigative Site, Cincinnati, Ohio
  - aTyr Investigative Site, Cleveland, Ohio
  - aTyr Investigative Site, Oklahoma City, Oklahoma
  - aTyr Investigative Site, Portland, Oregon
  - aTyr Investigative Site, Philadelphia, Pennsylvania
  - aTyr Investigative Site, Charleston, South Carolina
  - aTyr Investigative Site, Dickson, Tennessee
  - aTyr Investigative Site, Dallas, Texas
  - aTyr Investigative Site, Houston, Texas
  - aTyr Investigative Site, Salt Lake City, Utah
  - aTyr Investigative Site, Falls Church, Virginia
  - aTyr Investigative Site, Richmond, Virginia
- Brazil (4):
  - aTyr Investigative Site, Salvador, Estado de Bahia
  - aTyr Investigative Site, Porto Alegre, Rio Grande do Sul
  - aTyr Investigative Site, São Bernardo do Campo
  - aTyr Investigative Site, São Paulo
- France (5):
  - aTyr Investigative Site, Bobigny
  - aTyr Investigative Site, La Tronche
  - aTyr Investigative Site, Montpellier
  - aTyr Investigative Site, Paris
  - aTyr Investigative Site, Toulouse
- Germany (4):
  - aTyr Investigative Site, Essen
  - aTyr Investigative Site, Freiburg im Breisgau
  - aTyr Investigative Site, Hanover
  - aTyr Investigative Site, Heidelberg
- Italy (9):
  - aTyr Investigative Site, Catania
  - aTyr Investigative Site, Florence
  - aTyr Investigative Site, Forlì
  - aTyr Investigative Site, Milan
  - aTyr Investigative Site, Napoli
  - aTyr Investigative Site, Padua
  - aTyr Investigative Site, Rome
  - aTyr Investigative Site, Siena
  - aTyr Investigative Site, Trieste
- Japan (13):
  - Kyorin Investigative Site, Aomori
  - Kyorin Investigative Site, Fukuoka
  - Kyorin Investigative Site, Fukushima
  - Kyorin Investigative Site, Hokkaido
  - Kyorin Investigative Site, Hyōgo
  - Kyorin Investigative Site, Kanagawa
  - aTyr Investigative Site, Kumamoto
  - Kyorin Investigative Site, Miyagi
  - Kyorin Investigative Site, Okayama
  - Kyorin Investigative Site, Osaka
  - Kyorin Investigative Site, Shimane
  - Kyorin Investigative Site, Shizuoka
  - Kyorin Investigative Site, Tokyo
- aTyr Investigative Site, Nieuwegein, Netherlands
- Spain (4):
  - aTyr Investigative Site, Barcelona
  - aTyr Investigative Site, Madrid
  - aTyr Investigative Site, Santander
  - aTyr Investigative Site, Valencia
- United Kingdom (5):
  - aTyr Investigative Site, Birmingham
  - aTyr Investigative Site, Cambridge
  - aTyr Investigative Site, Cottingham
  - aTyr Investigative Site, Coventry
  - aTyr Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Forster S, Chong YE, Siefker D, Becker Y, Bao R, Escobedo E, Qing Y, Rauch K, Burman L, Burkart C, Kainz P, Cubitt A, Muders M, Nangle LA. Development and Characterization of a Novel Neuropilin-2 Antibody for Immunohistochemical Staining of Cancer and Sarcoidosis Tissue Samples. Monoclon Antib Immunodiagn Immunother. 2023 Oct;42(5):157-165. doi: 10.1089/mab.2023.0007. PMID 37902990